CLINICAL TRIAL: NCT02851511
Title: Augmenting Cognitive Training In Older Adults
Acronym: ACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: University of Arizona (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB201600785-N-R; R01AG054077 (NIH); RF1AG071469 (NIH); AWD00532 (Other: UFIRST)
Record Dates: First submitted 2016-07-07; First posted 2016-08-01 (Estimated); Results first posted 2023-07-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2023-06

CONDITIONS: Aging
MeSH Terms: interventions — Cognitive Training; Transcranial Direct Current Stimulation; Training Support

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Cognitive Training + Active Stimulation (Experimental): This arm receives cognitive training combined with active tDCS.
  Interventions: Behavioral: Cognitive Training; Device: tDCS (active stimulation)
- Cognitive Training + Sham Stimulation (Experimental): This arm receives cognitive training combined with sham tDCS.
  Interventions: Behavioral: Cognitive Training; Device: tDCS (sham stimulation)
- Educational Training + Active Stimulation (Experimental): This arm receives educational training combined with active tDCS.
  Interventions: Device: tDCS (active stimulation); Behavioral: Educational Training
- Educational Training + Sham Stimulation (Experimental): This arm receives educational training combined with sham tDCS.
  Interventions: Device: tDCS (sham stimulation); Behavioral: Educational Training

INTERVENTIONS:
Behavioral: Cognitive Training — Cognitive Training employs an eight component, PositScience BrainHQ suite via its researcher portal.
  Arms: Cognitive Training + Active Stimulation; Cognitive Training + Sham Stimulation
Device: tDCS (active stimulation) — A Soterix Clinical Trials Direct Current Stimulator will apply 20 minutes of 2.0mA direct current through two biocarbon rubber electrodes encased in saline soaked 5cm x 7cm sponges (8cc of 0.9% saline solution per sponge) placed over the frontal cortices at F3 and F4 (10-20 system).
  Arms: Cognitive Training + Active Stimulation; Educational Training + Active Stimulation
Device: tDCS (sham stimulation) — Sham stimulation is performed with the same device and all procedures will be identical except for the duration of stimulation. Participants will receive 30 seconds of 2 mA of direct current stimulation at the beginning of the session. Participants habituate to the sensation of tDCS within 30-60 seconds of stimulation. This procedure provides the same sensation of tDCS without the full duration of stimulation, making it a highly effective sham procedure.
  Arms: Cognitive Training + Sham Stimulation; Educational Training + Sham Stimulation
Behavioral: Educational Training — Educational training involves watching educational videos produced by the National Geographic Channel, which cover a range of topics such as history, nature, and wildlife. Participants will be asked to complete questions on the content of the videos to ensure sustained attention.
  Arms: Educational Training + Active Stimulation; Educational Training + Sham Stimulation

SUMMARY:
A two-phase adaptive randomized clinical trial will examine the individual and combined impact of pairing cognitive training with transcranial direct current stimulation (tDCS). tDCS is a method of non-invasive brain stimulation that directly stimulates brain regions involved in active cognitive function and could enhance neural plasticity when paired with a training task. We will compare changes in cognitive and brain function resulting from CT and ET combined with tDCS using a comprehensive neurocognitive, clinical, and multimodal neuroimaging assessment of brain structure, function, and metabolic state. Functional magnetic resonance imaging (FMRI) will be used to assess brain response during working memory, attention, and memory encoding; the active cognitive abilities trained by CT. Proton magnetic resonance spectroscopy (MRS) will assess cerebral metabolites, including GABA concentrations sensitive to neural plasticity. We hypothesize that: 1) tDCS will enhance neurocognitive function, brain function, and functional outcomes from CT, with combined CT and tDCS providing the most benefit; 2) Effects of tDCS on CT will be maintained up to 12 months following training, and 3) Neuroimaging biomarkers of cerebral metabolism, neural plasticity (GABA concentrations) and functional brain response (FMRI) during resting vs. active cognitive tasks will predict individual response to tDCS.

ELIGIBILITY:
Inclusion criteria:

1. Age 65 to 89 years; this age group was selected because it is at high risk of age-related cognitive decline and have a sufficiently long life expectancy to participate in the study.
2. Evidence of age-related cognitive decline in the Cognitive Training assessment defined by performance below the 80th percentile.
3. Ability to participate in the intervention and attend training sessions; willingness to be randomized to either treatment group.

Exclusion criteria:

1. Neurological disorders (e.g., dementia, stroke, seizures, traumatic brain injury).
2. Evidence of cognitive impairment (as defined by NACC UDS performance below 1.5 standard deviations on age/sex/education normative data in at least one cognitive domain).
3. Past opportunistic brain infection.
4. Major psychiatric illness (schizophrenia, intractable affective disorder, current substance dependence diagnosis or severe major depression and/or suicidality.
5. Unstable (e.g., cancer other than basal cell skin) and chronic (e.g. severe diabetes) medical conditions.
6. MRI contraindications (e.g., claustrophobia, metal implants).
7. Physical impairment precluding motor response or lying still for 1 hr and inability to walk two blocks without stopping.
8. Currently on GABA-ergic or glutamatergic medications, or on sodium channel blockers.
9. Left-handedness.

Ages: 65 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 379 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Woods, Ph.D, Principal Investigator — University of Florida
Locations (3):
- United States (3):
  - University of Arizona, Tucson, Arizona
  - Village of Gainesville, Gainesville, Florida
  - University of Florida McKnight Brain Institute, Gainesville, Florida

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant flow is reported with three periods. Period 1 includes all randomized participants (combined Phase I and Phase II). Period 2 contains only the Phase I participants. Period 3 contains only the Phase II participants.
  In Phase II the two education training arms were eliminated, hence the allocation of 0 to those groups. Participants who were enrolled in Phase I education training were not randomized again in Phase II (there is no crossover).
Period: Overall (Phase I + Phase II)
Arm/Group | Cognitive Training + Active Stimulation | Cognitive Training + Sham Stimulation | Educational Training + Active Stimulation | Educational Training + Sham Stimulation
Started | 168 | 166 | 23 | 22
Completed | 126 | 127 | 23 | 18
Not Completed | 42 | 39 | 0 | 4
Not completed — Physician Decision | 18 | 16 | 0 | 1
Not completed — Withdrawal by Subject | 20 | 17 | 0 | 3
Not completed — COVID-19 lockdown, no reason specified | 4 | 5 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Period: Phase I
Arm/Group | Cognitive Training + Active Stimulation | Cognitive Training + Sham Stimulation | Educational Training + Active Stimulation | Educational Training + Sham Stimulation
Started | 21 | 21 | 23 | 22
Completed | 19 | 20 | 23 | 18
Not Completed | 2 | 1 | 0 | 4
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 3
Period: Phase II
Arm/Group | Cognitive Training + Active Stimulation | Cognitive Training + Sham Stimulation | Educational Training + Active Stimulation | Educational Training + Sham Stimulation
Started | 147 | 145 | 0 | 0
Completed | 107 | 107 | 0 | 0
Not Completed | 40 | 38 | 0 | 0
Not completed — Physician Decision | 18 | 16 | 0 | 0
Not completed — Withdrawal by Subject | 18 | 16 | 0 | 0
Not completed — COVID-19 lockdown, no reason specified | 4 | 5 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study is a 2-phase adaptive design study. After first phase, 2 education arms were dropped. all participants were randomly assigned to 2 cognitive training groups in Phase II.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Training + Active Stimulation | Cognitive Training + Sham Stimulation | Educational Training + Active Stimulation | Educational Training + Sham Stimulation | Total
Number analyzed (Participants) | 168 | 166 | 23 | 22 | 379
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.5 (5.4) | 71.5 (4.8) | 70.0 (5.1) | 73.1 (4.7) | 71.5 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 111 | 10 | 11 | 236
  Male | 64 | 55 | 13 | 11 | 143
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 8 | 1 | 2 | 25
  Not Hispanic or Latino | 154 | 158 | 22 | 20 | 354
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 5 | 1 | 0 | 9
  Asian | 0 | 3 | 1 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  Black or African American | 11 | 8 | 0 | 2 | 21
  White | 146 | 148 | 20 | 18 | 332
  More than one race | 5 | 2 | 0 | 2 | 9
  Unknown or Not Reported | 3 | 0 | 0 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 168 | 166 | 23 | 22 | 0
Years of Education [Mean (Standard Deviation); unit: years] | 16.3 (2.3) | 16.4 (2.4) | 16.7 (2.1) | 15.6 (2.4) | 16.3 (2.4)
MOCA Total Score [Mean (Standard Deviation); unit: units on a scale] — Montreal Cognitive Assessment (MOCA) was designed as a rapid screening instrument for the detection of mild cognitive impairment. Higher scores indicate better cognition. The possible range of scores is 0 to 30. The total score is calculated by summing scores from the following domains: visuospatial/executive, naming, attention, language, abstraction, delayed recall, and orientation.
  units on a scale | 26.7 (2.0) | 26.8 (1.9) | 26.9 (1.7) | 26.1 (2.1) | 26.7 (1.9)
Average POSIT z-score: [Mean (Standard Deviation); unit: z-score] — POSIT BrainHQ Cognitive Training Composite Performance Measure (POSIT Z-Score) involves performance on the 8 selected cognitive training tasks set to the medium difficulty level and provides a measure of proximal performance on cognitive training tasks central to the cognitive training condition. A value of 0 represents mean performance as expected by age normative data. Higher positive values represent better than expected cognitive performance.
  z-score | -0.18 (0.44) | -0.20 (0.46) | -0.11 (0.47) | -0.44 (0.55) | -0.20 (0.46)
BDI-II Total Score [Mean (Standard Deviation); unit: units on a scale] — Beck Depression Inventory-II (BDI-II) measures the severity of depression in adolescents and adults. The total score ranges from 0 to 63 with higher scores indicating more severe depressive symptoms. Scores from 21 individual items are summed to create a total score.
  units on a scale | 4.0 (4.8) | 3.4 (3.9) | 2.4 (3.1) | 3.1 (3.7) | 3.6 (4.3)

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Cognitive Ability.
Description: Composite measure of cognitive ability as defined by NIH toolbox fluid cognition fully corrected T-score. Minimum change = -13, Maximum change = 26. Higher scores mean a better outcome. The minimum and maximum for Cognitive Training + Active Stimulation, Cognitive Training + Sham Stimulation, Educational Training + Active Stimulation and Educational Training + Sham Stimulation are (-13, 20) and (-10, 26), respectively. This outcome is measured for the participants who received cognitive training, including both Phase I and Phase II participants, N=334 (Phase I N=42, Phase II N=292).
Time Frame: Change from baseline to post assessment (3 months).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Training + Active Stimulation | Cognitive Training + Sham Stimulation
Number analyzed (Participants) | 168 | 166
units on a scale | 4.7 (6.5) | 4.5 (6.1)
Statistical Analysis 1: Comparison: Cognitive Training + Active Stimulation vs Cognitive Training + Sham Stimulation; Null hypothesis: The combination of cognitive training (12 weeks) and active stimulation (over the dorsolateral prefrontal cortex) will not lead to beneficial changes on the NIH Toolbox Cognition Battery. The study is designed to have at least 90% power to detect a difference of effect size 0.42 between cognitive training+tDCS and cognitive training+sham, using a normal inverse combination test at one-sided 0.025 level; Test type: Superiority — tDCS vs. sham superiority with cognitive training will be tested based on the 320 participants who are assigned to the two cognitive training arms. The effects of tDCS on changes in NIH Toolbox Fluid Cognition Composite Score (NIHTB FCC) from baseline to 3-month follow-up are estimated by linear regression models, with missing outcomes predicted by regression models that include demographic and baseline characteristics; p < 0.05, Regression, Linear — Formal statistical inference of the tDCS effect was based on the inverse-normal combination of two p-values, one from the Phase I data (N=42) and the other from the Phase II data (N=292); Slope = 0.33, 95% CI 2-sided [-0.91 to 1.56], Standard Error of Mean 0.63

2. Secondary Outcome: Phase I POSIT BrainHQ Cognitive Training Composite Performance Measure.(Phase I POSIT Z-Score)
Description: POSIT BrainHQ Cognitive Training Composite Performance measure involves performance on the 8 selected cognitive training tasks set to the medium difficulty level and provides a measure of proximal performance on cognitive training tasks central to the cognitive training condition. The higher score indicates better performance. The range of POSIT Z-Score at 3-month is -1.04 to 1.75. the minimum and maximum for Cognitive training group and Education training group are (-0.24, 1.75) and (-1.04, 1.39), respectively.
Time Frame: Baseline to post assessment (3 months).
Population: Adults were between the ages of 65-89, right-handed, fluent in English, and had evidence of age-related cognitive decline. Analysis includes all 87 participants from Phase I.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Cognitive Training: This arm receives cognitive training.
  Cognitive Training: Cognitive Training employs an eight component, PositScience BrainHQ suite via its researcher portal.
- Education Training: This arm receives education training.
  Educational Training: Educational training involves watching educational videos produced by the National Geographic Channel, which cover a range of topics such as history, nature, and wildlife. Participants will be asked to complete questions on the content of the videos to ensure sustained attention.
Arm/Group | Cognitive Training | Education Training
Number analyzed (Participants) | 42 | 45
units on a scale | 0.95 (0.41) | -0.06 (0.47)

ADVERSE EVENTS:
Time Frame: The adverse events were collected over an approximate one year period. They were collected from study enrollment until the 1 year followup visit.
Description: Adverse events were queried using medical history questionnaires at baseline, 3 month post test, and 1 follow-up assessment visits. If adverse events were self reported by participants between assessment visits a standardized adverse event form was completed to assess severity, relatedness, and outcome.
Arm/Group | Cognitive Training + Active Stimulation | Cognitive Training + Sham Stimulation | Educational Training + Active Stimulation | Educational Training + Sham Stimulation
All-Cause Mortality (participants affected / at risk) | 0/168 | 0/166 | 0/23 | 0/22
Serious Adverse Events (participants affected / at risk) | 16/168 | 19/166 | 4/23 | 5/22
Other Adverse Events (participants affected / at risk) | 69/168 | 75/166 | 12/23 | 12/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive Training + Active Stimulation (N=168) | Cognitive Training + Sham Stimulation (N=166) | Educational Training + Active Stimulation (N=23) | Educational Training + Sham Stimulation (N=22)
Accidentally swallowed non food item (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Allergic reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anterior and posterior surgery (pelvic floor) (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bleeding (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood Loss (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bowel Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bowel infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Broken finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cat bite (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest Pain (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Cut on cheek (stiches) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cyst removal (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dislocated Shoulder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Esophageal cancer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye injury (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (General disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Fall (fractured finger) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fecal blockage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Finger injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foot fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herniated disc repair (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection from Knee Replacement (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection from skin wound (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal Bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate Cancer (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rapid heartbeat (ER visit) (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Shingles (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Shortness of Breath, tunnel vision, lost continence (ER visit) (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin cancer spot removal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Stitches (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomach bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Torn artery (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transient ischemic attack (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urine retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive Training + Active Stimulation (N=168) | Cognitive Training + Sham Stimulation (N=166) | Educational Training + Active Stimulation (N=23) | Educational Training + Sham Stimulation (N=22)
Actinic Keratoses (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anxiety and Depression (Psychiatric disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 8 (12) | 8 (10) | 0 (0) | 2 (2)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (urgent care visit) (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Bipolar Disorder Treatment (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bladder infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Bone fusion of finger (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone spur (foot) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone spurs on knees (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast Cancer (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Broken bone in hand from fall (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Broken wrist (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bruised rib (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cataract surgery (Surgical and medical procedures) | 10 (11) | 6 (7) | 1 (1) | 0 (0)
Cataracts (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest Pain (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (caused by esophogeal gastritis and hiatal hernia) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colonoscopy (Surgical and medical procedures) | 3 (3) | 2 (2) | 0 (0) | 1 (1)
Concussion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough / Allergies (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cut on head (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Dizziness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enlarged prostate (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye hemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye injury (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eyelid surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fainting (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fainting (post blood draw unrelated to study) (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Fall (hit front of head) (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Finger numbness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Foot Injury (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Fractured hand (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hearing impairment (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hearing loss (Ear and labyrinth disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Heart Ablation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heart Murmur (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heart palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Heat Exhaustion (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hernia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
High Blood Pressure (Cardiac disorders) | 6 (6) | 1 (1) | 0 (0) | 1 (1)
High Cholesterol (General disorders) | 3 (3) | 7 (7) | 0 (0) | 0 (0)
High blood pressure and low heart rate (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hip Replacement (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hip injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Kidney Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Kidney stones (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Knee Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Knee and hip pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Knee injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Larynopharyngeal reflux (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Low Iron (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Macular degeneration (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Migraine headache (Nervous system disorders) | 6 (9) | 10 (14) | 1 (1) | 1 (1)
Mononucleosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal Drip (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nausea and Dizziness (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Neck Injury from car accident (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral surgery (Surgical and medical procedures) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
PTSD & Increased Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paronychia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Posterior Vitreous Detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Protruding Disc (L5) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Radio ablation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Shingles (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin biopsy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin cancer spot removal (Surgical and medical procedures) | 19 (23) | 24 (31) | 4 (5) | 3 (4)
Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal Stenosis & Sciatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stents (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stress fracture (fibula) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sty (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thoracic Aortic Aneurysm (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 3 (3) | 9 (10) | 1 (3) | 3 (3)
Urolift implant (Enlarged Prostate treatment) (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Varithena Ablation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Varithena treatment (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Nervous system disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Wrist pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wrist surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-16): https://cdn.clinicaltrials.gov/large-docs/11/NCT02851511/Prot_SAP_000.pdf
  • Informed Consent Form (2019-02-11): https://cdn.clinicaltrials.gov/large-docs/11/NCT02851511/ICF_001.pdf